CLINICAL TRIAL: NCT03083938
Title: Prospective Randomized Controlled Trial of Omental Roll-up Technique on Pancreato-jejunostomy Anastomosis for Reducing Perioperative Complication in Patients Undergoing Pancreatoduodenectomy
Brief Title: Trial of Omental Roll-up Technique on Pancreato-jejunostomy Anastomosis for Reducing Perioperative Complication in Patients Undergoing Pancreatoduodenectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Paramin Muangkaew, MD, Principal Investigator, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ID 12-59-13
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2017-08-29 (Actual); Status verified 2017-08

CONDITIONS: Periampullary Carcinoma; Pancreatic Fistula
Keywords: Pancreatoduodenectomy; Omentum; Wrapping; Roll-up; Whipple
MeSH Terms: conditions — Pancreatic Fistula

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Omental Roll-up (Experimental)
  Interventions: Procedure: Omental Roll-up
- No Omental Roll-up (No Intervention)

INTERVENTIONS:
Procedure: Omental Roll-up — Using omentum roll-up pancreato-jejunal anastomosis
  Arms: Omental Roll-up

SUMMARY:
Despite the fact that pancreatoduodenectomy is the standard treatment of malignant tumor at periampullary area, the morbidity and mortality rate with intra-abdominal collection, post pancreatectomy hemorrhage, and delayed gastric emptying, is still high at approximately 50-60%. The causes of these complications usually come from post-operative pancreatic fistula. Nowadays, several methods have been reported to reduce the incidence of pancreatic fistula after undergoing pancreatoduodenectomy, such as pancreatic stenting, the use of intravenous somatostatin, the use of sealant material and wrapping anastomosis by soft tissue.

Wrapping pancreato-jejunal anastomosis with omentum is not a complicate procedure and requires no extra treatment expenses of the patient. It has been reported this technique has been applied in the non-randomized controlled trials and their data have significantly shown that the technique could reduce pancreatic fistula rate. Therefore, the researchers want to conduct an RCT study to compare complication rates between omental roll-up pancreato-jejunal anastomosis and non-omental roll-up groups.

DETAILED DESCRIPTION:
This is a RCT study designed to compare the use of omental roll-up technique with non-omental roll-up technique at pancreato-jejunal anastomosis in patients undergoing pancreatoduodenectomy. The purpose of this study is to prove the hypothesis that omental roll-up technique can reduce the complication rate or pancratic fistula after pancreatoduodenectomy. This study was approved by the committee on human rights to conduct the research involving human subjects, faculty of medicine Ramathibodi hospital, Mahidol university. The patients are operated by experienced surgeons of Hepato-pancreato-biliary unit, department of surgery, Ramathibodi hospital and randomized into two groups by using the closed envelope method after completing pancreato-jejunal anastomosis. Then, patients are followed-up and the data are collected for 30 days after the surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing pancreatoduodenectomy from these disease, carcinoma at head of pancreas, carcinoma at ampullar of Vater, Distal cholangiocarcinoma, Carcinoma of duodenum

Exclusion Criteria:

* Unresectable pancreatoduodenectomy
* Patients underwent omentectomy from prior surgery

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-04-01 (Estimated); Study Completion 2019-05-01 (Estimated)

PRIMARY OUTCOMES:
Complication rate after using omental roll-up technique | Within 30 days after surgery
  Complication rate after using omental roll-up technique compare with non-omental roll-up

SECONDARY OUTCOMES:
Pancreatic fistula rate after using omental roll-up technique | Within 30 days after surgery
  Pancreatic fistula rate after using omental roll-up technique compare with non-omental roll-up

CONTACTS AND LOCATIONS:
Locations (1):
- Paramin Muangkaew, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sakamoto Y, Shimada K, Esaki M, Kajiwara T, Sano T, Kosuge T. Wrapping the stump of the gastroduodenal artery using the falciform ligament during pancreaticoduodenectomy. J Am Coll Surg. 2007 Feb;204(2):334-6. doi: 10.1016/j.jamcollsurg.2006.11.015. No abstract available. PMID 17254940
- [Background] Iannitti DA, Coburn NG, Somberg J, Ryder BA, Monchik J, Cioffi WG. Use of the round ligament of the liver to decrease pancreatic fistulas: a novel technique. J Am Coll Surg. 2006 Dec;203(6):857-64. doi: 10.1016/j.jamcollsurg.2006.08.021. Epub 2006 Oct 25. PMID 17116554
- [Background] Ramia JM, de la Plaza R, Adel F, Ramiro C, Arteaga V, Garcia-Parreno J. Wrapping in pancreatic surgery: a systematic review. ANZ J Surg. 2014 Dec;84(12):921-4. doi: 10.1111/ans.12491. Epub 2013 Dec 19. PMID 25720806
- [Background] Choi SB, Lee JS, Kim WB, Song TJ, Suh SO, Choi SY. Efficacy of the omental roll-up technique in pancreaticojejunostomy as a strategy to prevent pancreatic fistula after pancreaticoduodenectomy. Arch Surg. 2012 Feb;147(2):145-50. doi: 10.1001/archsurg.2011.865. PMID 22351908